CLINICAL TRIAL: NCT01168856
Title: A Long-term Monitoring Study to Evaluate the Persistence of Direct Antiviral (DAA) Treatment Resistant Mutations or the Durability of Sustained Virological Response (SVR) in Patients Treated With DAA Containing Regimens for Chronic Hepatitis C Infections (CHC)
Brief Title: An Observational Study on Long-Term Persistence of Resistant Mutations And Durability of Sustained Virological Response in Patients With Chronic Hepatitis C Treated With Direct Acting Antiviral (DAA)- Containing Regimens
Status: Terminated | Type: Observational
Why Stopped: This study was terminated due to the decrease in percentage of participants.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: NV22688; 2009-016560-36 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-23 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum specimens collected from patients with partial viral response or viral load rebound of viral response to monitor for resistance mutations in viral RNA

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational long-term follow-up study will assess the persistence of direct acting antiviral (DAA) resistant mutations and the durability of sustained virological response in patients with chronic hepatitis C who have participated in a Roche DAA treatment protocol. Up to 5 scheduled monitoring visits for blood sampling during an observational period of up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* chronic hepatitis C
* participation in Roche DAA treatment protocol for CHC infection
* DAA-associated resistant mutations persisting through to last evaluation in donor protocol , or partial viral response or viral load rebound while on RO5024048 treatment, or sustained virological response >/= 20 weeks after last dose of study medication in donor study

Exclusion Criteria:

* For patients participating in DAA resistance monitoring: Initiation of treatment after participation in the donor protocol for which there is evidence of cross-resistance to donor protocol DAA
* For patients participating in DAA SVR durability: Treatment with any anti-HVC therapy since establishing SVR in the donor study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C patients having received direct acting antiviral treatment in donor protocol
Sampling Method: Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2010-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (104):
- United States (31):
  - La Jolla, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Bradenton, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Hillsborough, New Jersey
  - Newark, New Jersey
  - Manhasset, New York
  - New York, New York
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Newport News, Virginia
  - Richmond, Virginia
  - Vancouver, Washington
- Australia (9):
  - Darlinghurst, New South Wales
  - Kingswood, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - Greenslopes, Queensland
  - Herston, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Melbourne, Victoria
- Vienna, Austria
- Brazil (3):
  - Salvador, Estado de Bahia
  - Porto Alegre, Rio Grande do Sul
  - Ribeirão Preto, São Paulo
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (11):
  - Clichy
  - Créteil
  - Lille
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Rennes
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (5):
  - Berlin
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - München
- Italy (7):
  - Bari, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Milan, Lombardy
  - Pavia, Lombardy
  - Turin, Piedmont
  - Pisa, Tuscany
- Mexico (2):
  - Guadalajara
  - Monterrey
- New Zealand (3):
  - Christchurch
  - Dunedin
  - Grafton
- Poland (6):
  - Bydgoszcz
  - Chorzów
  - Lodz
  - Mysłowice
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Bratislava, Slovakia
- Spain (10):
  - Palma de Mallorca, Balearic Islands
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Santander, Cantabria
  - A Coruña, La Coruña
  - Madrid, Madrid
  - Pontevedra, Pontevedra
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia
- United Kingdom (5):
  - Dorset
  - Dundee
  - London
  - Manchester
  - Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from following studies were enrolled: NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094].
Pre-assignment Details: This study was terminated early and participants discontinued due to study termination were included under reason "unspecified" in the participant flow.
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with Hepatitis C Virus (HCV) infection who participated in one of the following studies (Donor Protocols: NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094]) and had developed direct acting antiviral (DAA)-associated resistant mutation(s), which persisted through to the last evaluation of drug resistance in the donor protocol(s), or achieved only a partial viral response or experienced a viral breakthrough while on mericitabine treatment not associated with selection of S282T resistance mutations. Participants were monitored up to 18 months.
- Sustained Virological Response (SVR) Durability Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following studies (NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094]) and had achieved Sustained Virological Response (SVR), defined within the donor protocol as measured by the Roche COBAS TaqMan HCV Test greater than or equal to (≥) 20 weeks after the last dose of study medication. Participants were monitored up to 36 months.
Period: Overall Study
Arm/Group | Resistance Monitoring Arm | Sustained Virological Response (SVR) Durability Monitoring Arm
Started | 176 | 558
Completed | 158 | 215
Not Completed | 18 | 343
Not completed — Lost to Follow-up | 4 | 34
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Physician Decision | 2 | 1
Not completed — Confirmed Quantifiable HCV RNA | 0 | 1
Not completed — Participant received anti-HCV treatment | 1 | 0
Not completed — Death | 0 | 2
Not completed — Other | 1 | 291
Not completed — Protocol Violation | 4 | 6

BASELINE CHARACTERISTICS:
Population: Eligible population included all enrolled participants excluding participants with protocol violations.
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following studies (Donor Protocols: NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094]) and had developed DAA-associated resistant mutation(s), which persisted through to the last evaluation of drug resistance in the donor protocol(s), or achieved only a partial viral response or experienced a viral breakthrough while on mericitabine treatment not associated with selection of S282T resistance mutations. Participants were monitored up to 18 months.
- SVR Durability Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following studies (NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094]) and had achieved SVR, defined within the donor protocol as measured by the Roche COBAS TaqMan HCV Test ≥ 20 weeks after the last dose of study medication. Participants were monitored up to 36 months.
- Total: Total of all reporting groups
Arm/Group | Resistance Monitoring Arm | SVR Durability Monitoring Arm | Total
Number analyzed (Participants) | 172 | 552 | 724
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (8.48) | 51.0 (10.79) | 51.2 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 222 | 269
  Male | 125 | 330 | 455

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With the Detectable HCV Ribonucleic Acid (RNA) Results in Resistance Monitoring Arm at Month 3
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 International Units per milliliter [IU/mL]).
Time Frame: Month 3
Population: Resistance monitoring population included all participants who were enrolled in resistance monitoring arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 3.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 114
Percentage of participants | 99.1

2. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in Resistance Monitoring Arm at Month 6
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 6
Population: Resistance monitoring population included all participants who were enrolled in resistance monitoring arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 6.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 137
Percentage of participants | 99.3

3. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in Resistance Monitoring Arm at Month 9
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 9
Population: Resistance monitoring population included all participants who were enrolled in resistance monitoring arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 129
Percentage of participants | 99.2

4. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in Resistance Monitoring Arm at Month 12
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 12
Population: Resistance monitoring population included all participants who were enrolled in resistance monitoring arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 123
Percentage of participants | 99.2

5. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in Resistance Monitoring Arm at Month 18
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 18
Population: Resistance monitoring population included all participants who were enrolled in resistance monitoring arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 18.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 113
Percentage of participants | 100

6. Primary Outcome: HCV RNA Levels in Resistance Monitoring Arm at Month 3
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 3
Population: Resistance monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 3.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 113
IU/mL | 3922296 (5111469)

7. Primary Outcome: HCV RNA Levels in Resistance Monitoring Arm at Month 6
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 6
Population: Resistance monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 6.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 136
IU/mL | 4369148 (6803658)

8. Primary Outcome: HCV RNA Levels in Resistance Monitoring Arm at Month 9
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 9
Population: Resistance monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 9.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 128
IU/mL | 5016299 (7235510)

9. Primary Outcome: HCV RNA Levels in Resistance Monitoring Arm at Month 12
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 12
Population: Resistance monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 12.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 122
IU/mL | 4955311 (6595493)

10. Primary Outcome: HCV RNA Levels in Resistance Monitoring Arm at Month 18
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 18
Population: Resistance monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 18.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 113
IU/mL | 4830852 (6621059)

11. Primary Outcome: Mean Systolic Blood Pressure in Resistance Monitoring Arm at Month 3
Description: Any abnormalities in systolic blood pressure (units: millimeters of Mercury [Hg] [mmHg]) were reported at the discretion of principal investigator.
Time Frame: Month 3
Population: Resistance monitoring population. Here, number of participants analyzed = participants with vital signs assessment at Month 3.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 111
mmHg | 128.1 (16.15)

12. Primary Outcome: Systolic Blood Pressure in Resistance Monitoring Arm at Month 6
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 6
Population: Resistance monitoring population. Here, number of participants analyzed = participants with vital signs assessment at Month 6.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 134
mmHg | 126.0 (16.58)

13. Primary Outcome: Systolic Blood Pressure in Resistance Monitoring Arm at Month 9
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 9
Population: Resistance monitoring population. Here, number of participants analyzed = participants with vital signs assessment at Month 9.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 128
mmHg | 126.9 (15.48)

14. Primary Outcome: Mean Systolic Blood Pressure in Resistance Monitoring Arm at Month 12
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 12
Population: Resistance monitoring population. Here, number of participants analyzed = participants with vital signs assessment at Month 12.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 122
mmHg | 127.1 (14.97)

15. Primary Outcome: Mean Systolic Blood Pressure in Resistance Monitoring Arm at Month 18
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 18
Population: Resistance monitoring population. Here, number of participants analyzed = participants with vital signs assessment at Month 18.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 114
mmHg | 130.3 (17.53)

16. Primary Outcome: Mean Diastolic Blood Pressure in Resistance Monitoring Arm at Month 3
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 111
mmHg | 79.8 (10.67)

17. Primary Outcome: Mean Diastolic Blood Pressure in Resistance Monitoring Arm at Month 6
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 134
mmHg | 78.0 (10.60)

18. Primary Outcome: Mean Diastolic Blood Pressure in Resistance Monitoring Arm at Month 9
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 9
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 128
mmHg | 78.5 (9.60)

19. Primary Outcome: Mean Diastolic Blood Pressure in Resistance Monitoring Arm at Month 12
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 122
mmHg | 77.7 (9.92)

20. Primary Outcome: Mean Diastolic Blood Pressure in Resistance Monitoring Arm at Month 18
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 18
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 114
mmHg | 79.3 (9.77)

21. Primary Outcome: Mean Pulse Rate in Resistance Monitoring Arm at Month 3
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 111
Beats per minute | 70.6 (9.89)

22. Primary Outcome: Mean Pulse Rate in Resistance Monitoring Arm at Month 6
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 134
Beats per minute | 71.1 (10.14)

23. Primary Outcome: Mean Pulse Rate in Resistance Monitoring Arm at Month 9
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 9
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 128
Beats per minute | 70.3 (12.08)

24. Primary Outcome: Mean Pulse Rate in Resistance Monitoring Arm at Month 12
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 122
Beats per minute | 70.3 (10.68)

25. Primary Outcome: Mean Pulse Rate in Resistance Monitoring Arm at Month 18
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 18
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 114
Beats per minute | 70.8 (10.75)

26. Primary Outcome: Percentage of Participants Who Received Anti-HCV Medications in Resistance Monitoring Arm
Description: Percentage of participants who received any anti-HCV medication during the monitoring period was reported.
Time Frame: Up to 18 months
Population: Resistance monitoring population.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 172
Percentage of participants | 1.2

27. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in SVR Durability Monitoring Arm at Month 6
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 6
Population: SVR durability monitoring population included all participants who were enrolled in SVR durability arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 6.
Measure: Number; unit: Percentage of participants
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 505
Percentage of participants | 0.2

28. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in SVR Durability Monitoring Arm at Month 12
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 12
Population: SVR durability monitoring population included all participants who were enrolled in SVR durability arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 12.
Measure: Number; unit: Percentage of participants
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 516
Percentage of participants | 0

29. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in SVR Durability Monitoring Arm at Month 24
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 24
Population: SVR durability monitoring population included all participants who were enrolled in SVR durability arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 24.
Measure: Number; unit: Percentage of participants
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 416
Percentage of participants | 0

30. Primary Outcome: Percentage of Participants With the Detectable HCV RNA Results in SVR Durability Monitoring Arm at Month 36
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 36
Population: SVR durability monitoring population included all participants who were enrolled in SVR durability arm. Here, number of participants analyzed = participants with HCV RNA assessment at Month 36.
Measure: Number; unit: Percentage of participants
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 214
Percentage of participants | 0

31. Primary Outcome: Mean HCV RNA Levels in SVR Durability Monitoring Arm at Month 6
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 6
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 6.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 1
IU/mL | 896000

32. Primary Outcome: Mean HCV RNA Levels in SVR Durability Monitoring Arm at Month 12
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 12
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 12.
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 0

33. Primary Outcome: Mean HCV RNA Levels in SVR Durability Monitoring Arm at Month 24
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 24
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 24.
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 0

34. Primary Outcome: Mean HCV RNA Levels in SVR Durability Monitoring Arm at Month 36
Description: Serum HCV RNA concentration was determined using the Roche COBAS TaqMan HCV Test (Detection limit = 15 IU/mL).
Time Frame: Month 36
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with detectable HCV RNA at Month 36.
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 0

35. Primary Outcome: Mean Systolic Blood Pressure in SVR Durability Monitoring Arm at Month 6
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 6
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with vital signs assessments at Month 6.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 493
mmHg | 126.8 (16.83)

36. Primary Outcome: Mean Systolic Blood Pressure in SVR Durability Monitoring Arm at Month 12
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 12
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with vital signs assessments at Month 12.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 511
mmHg | 127.4 (16.66)

37. Primary Outcome: Mean Systolic Blood Pressure in SVR Durability Monitoring Arm at Month 24
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 24
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with vital signs assessments at Month 24.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 411
mmHg | 128.0 (15.56)

38. Primary Outcome: Mean Systolic Blood Pressure in SVR Durability Monitoring Arm at Month 36
Description: Any abnormalities in systolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 36
Population: SVR durability monitoring population. Here, number of participants analyzed = participants with vital signs assessments at Month 36.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 209
mmHg | 130.1 (16.68)

39. Primary Outcome: Mean Diastolic Blood Pressure in SVR Durability Monitoring Arm at Month 6
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 493
mmHg | 77.9 (10.67)

40. Primary Outcome: Mean Diastolic Blood Pressure in SVR Durability Monitoring Arm at Month 12
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 12
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 511
mmHg | 78.0 (10.31)

41. Primary Outcome: Mean Diastolic Blood Pressure in SVR Durability Monitoring Arm at Month 24
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 24
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 411
mmHg | 78.3 (10.28)

42. Primary Outcome: Mean Diastolic Blood Pressure in SVR Durability Monitoring Arm at Month 36
Description: Any abnormalities in diastolic blood pressure were reported at the discretion of principal investigator.
Time Frame: Month 36
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 209
mmHg | 78.3 (10.11)

43. Primary Outcome: Mean Pulse Rate in SVR Durability Monitoring Arm at Month 6
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 493
Beats per minute | 72.0 (10.41)

44. Primary Outcome: Mean Pulse Rate in SVR Durability Monitoring Arm at Month 12
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 12
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 511
Beats per minute | 72.9 (9.61)

45. Primary Outcome: Mean Pulse Rate in SVR Durability Monitoring Arm at Month 24
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 24
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 411
Beats per minute | 72.7 (10.45)

46. Primary Outcome: Mean Pulse Rate in SVR Durability Monitoring Arm at Month 36
Description: Any abnormalities in pulse rate were reported at the discretion of principal investigator.
Time Frame: Month 36
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | SVR Durability Monitoring Arm
Number analyzed (Participants) | 209
Beats per minute | 73.0 (11.10)

47. Primary Outcome: Number of Participants With Danoprevir (DNV) Resistance Status-Population Sequencing
Description: Population sequencing was used for determination of loss of resistance status. Resistance status was reported as either with loss of DNV resistance or without loss of DNV resistance.
  Results are reported as per donor protocol. Category 1: Number of participants with loss of resistance in NV22688. A total of 99 participants with resistance at the end of donor study by population sequencing were included in this analysis.
  Category 2: Number of participants with no loss of resistance in NV22688. A total of 33 participants with resistance at the end of donor study by population sequencing were included in this analysis.
  Category 3: Number of participants with loss of resistance in donor study. A total of 30 participants with no DNV resistance at the end of donor study by population sequencing enrolled in NV22688 were included in this analysis.
Time Frame: Month 3-18
Population: Resistance monitoring population.
Measure: Number; unit: participants
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following donor protocols: NV21075 [NCT00963885], WV21913 [NCT01331850], NP22660 [NCT01185860], NV22776 [NCT01220947], PP25213 [NCT01278134], NP27946 [NCT01483742], NP28266 [NCT01628094]. Patients had developed DNV-associated resistant mutation(s), which persisted or not through to the last evaluation of drug resistance in the donor protocol(s). Participants were monitored up to 18 months.
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 162
participants
  NP22660 Category 1 | 3
  NP22660 Category 2 | 0
  NP22660 Category 3 | 1
  NP27946 Category 1 | 1
  NP27946 Category 2 | 3
  NP27946 Category 3 | 1
  NV21075 Category 1 | 4
  NV21075 Category 2 | 1
  NV21075 Category 3 | 1
  NP28266 Category 1 | 4
  NP28266 Category 2 | 1
  NP28266 Category 3 | 6
  NV22776 Category 1 | 17
  NV22776 Category 2 | 6
  NV22776 Category 3 | 6
  PP25213 Category 1 | 37
  PP25213 Category 2 | 11
  PP25213 Category 3 | 1
  WV21913 Category 1 | 33
  WV21913 Category 2 | 11
  WV21913 Category 3 | 14

48. Primary Outcome: Number of Participants With DNV Resistance Status-Clonal Sequencing
Description: Clonal sequencing was used for determination of loss of resistance status. Resistance status was reported as either with loss of DNV resistance or without loss of DNV resistance.
  Category 1-Number of participants with loss of resistance in NV22688. A total of 64 participants with loss of resistance in NV22688 were included in this analysis.
  Category 2-Number of participants with no loss of resistance in NV22688. A total of 35 participants with no loss of resistance in NV22688 were included in this analysis.
  Category 3-Number of participants with loss of resistance in donor study. A total of 26 participants who had no DNV resistance at the end of donor study were analyzed by clonal sequencing in NV22688. Three participants from donor studies WV21913, NP28266 and NP27946, respectively were not analyzed by clonal sequencing in NV22688 as loss of resistance mutations was demonstrated by clonal sequencing in donor study.
Time Frame: Month 3-18
Population: Resistance monitoring population.
Measure: Number; unit: participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 125
participants
  NP27946 Category 1 | 1
  NP27946 Category 2 | 0
  NP27946 Category 3 | 0
  NP22660 Category 1 | 3
  NP22660 Category 2 | 0
  NP22660 Category 3 | 1
  NV21075 Category 1 | 2
  NV21075 Category 2 | 2
  NV21075 Category 3 | 1
  NP28266 Category 1 | 3
  NP28266 Category 2 | 1
  NP28266 Category 3 | 4
  NV22776 Category 1 | 9
  NV22776 Category 2 | 8
  NV22776 Category 3 | 6
  PP25213 Category 1 | 21
  PP25213 Category 2 | 16
  PP25213 Category 3 | 1
  WV21913 Category 1 | 25
  WV21913 Category 2 | 8
  WV21913 Category 3 | 13

49. Primary Outcome: Number of Participants With Boceprevir (BOC) or Telaprevir (TVR) Resistance Status-Population Sequencing
Description: Population sequencing was used for determination of loss of resistance status. Resistance status was reported as either with loss of BOC or TVR resistance or without loss of BOC or TVR resistance.
  Category 1-Number of participants with loss of resistance in NV22688. A total of 6 participants with resistance at the end of donor study by population sequencing were included in this analysis.
  Category 2-Number of participants with no loss resistance in NV22688. One participant with resistance at the end of donor study by population sequencing was included in this analysis.
  Category 3-Number of participants with loss of resistance in donor study. A total of 2 participants with no BOC or TVR resistance at the end of donor study by population sequencing enrolled in NV22688 were included in this analysis.
Time Frame: Month 3-18
Population: Resistance monitoring population.
Measure: Number; unit: participants
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following donor protocols: NV21075 [NCT00963885], WV21913 [NCT01331850], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NP27946 [NCT01483742], NP28266 [NCT01628094]. Patients had developed DNV-associated resistant mutation(s), which persisted or not through to the last evaluation of drug resistance in the donor protocol(s). Participants were monitored up to 18 months.
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 9
participants
  TVR study NV22779 Category 1 | 3
  TVR study NV22779 Category 2 | 1
  TVR study NV22779 Category 3 | 1
  BOC study NV22780 Category 1 | 3
  BOC study NV22780 Category 2 | 0
  BOC study NV22780 Category 3 | 1

50. Primary Outcome: Number of Participants With BOC or TVR Resistance Status-Clonal Sequencing
Description: Clonal sequencing was used for determination of loss of resistance status. Resistance status was reported as either with loss of BOC or TVR resistance or without loss of BOC or TVR resistance.
  Category 1-Number of participants with loss of resistance in NV22688. A total of 3 participants with loss of resistance in NV22688 were included in this analysis.
  Category 2-Number of participants with no loss of resistance in NV22688. A total of 3 participants with no loss of resistance in NV22688 were included in this analysis.
  Category 3-Number of participants with loss of resistance in donor study. A total of 2 participants who had no resistance at the end of donor study were analyzed by clonal sequencing in NV22688.
Time Frame: Month 3-18
Population: Resistance monitoring population.
Measure: Number; unit: participants
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following donor protocols: NV27779 [NCT01482390], NV27780 [NCT01482403]. Patients had developed BOC- or TVR-associated resistant mutation(s), which persisted or not through to the last evaluation of drug resistance in the donor protocol(s). Participants were monitored up to 18 months.
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 8
participants
  TVR study NV22779 Category 1 | 2
  TVR study NV22779 Category 2 | 1
  TVR study NV22779 Category 3 | 1
  BOC study NV22780 Category 1 | 1
  BOC study NV22780 Category 2 | 2
  BOC study NV22780 Category 3 | 1

51. Primary Outcome: Number of Participants With Setrobuvir (STV) Resistance Status-Population Sequencing
Description: Population sequencing was used for determination of loss of resistance status. Resistance status was reported as either with loss of STV resistance or without loss of STV resistance.
  Category 1-Number of participants with loss of resistance in NV22688. A total of 5 participants with resistance at the end of donor study by population sequencing were included in this analysis.
  Category 2-Number of participants with no loss resistance in NV22688. A total of 3 participants with resistance at the end of donor study by population sequencing were included in this analysis.
  Category 3-Number of participants with loss of resistance in donor study. A total of 3 participants with no STV resistance at the end of donor study by population sequencing enrolled in NV22688 were included in this analysis.
Time Frame: Month 3-18
Population: Resistance monitoring population.
Measure: Number; unit: participants
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in the following donor protocol: NP28266 [NCT01628094]. Patients had developed STV-associated resistant mutation(s), which persisted or not through to the last evaluation of drug resistance in the donor protocol(s). Participants were monitored up to 18 months.
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 11
participants
  NP28266 Category 1 | 5
  NP28266 Category 2 | 3
  NP28266 Category 3 | 3

52. Primary Outcome: Number of Participants With STV Resistance Status-Clonal Sequencing
Description: Clonal sequencing was used for determination of loss of resistance status. Resistance status was reported as either with loss of STV resistance or without loss of STV resistance.
  Category 1-Number of participants with loss of resistance in NV22688. One participant with loss of resistance in NV22688 was included in this analysis.
  Category 2-Number of participants with no loss of resistance in NV22688. A total of 4 participants with no loss of resistance in NV22688 were included in this analysis.
  Category 3-Number of participants with loss of resistance in donor study. One participant with loss of resistance, analyzed by clonal sequencing in NV22688.
  Category 4-Number of participants with loss of resistance in donor study. Two participants with no loss of resistance, analyzed by clonal sequencing in NV22688.
Time Frame: Month 3-18
Population: Resistance monitoring population. Here, n1=total number of participants with loss of STV resistance in NV22688 (by population sequencing). n2= total number of participants who had no STV resistance at the end of donor study they experienced a viral relapse in NV22688.
Measure: Number; unit: participants
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 8
participants
  NP28266 Category 1 | 1
  NP28266 Category 2 | 4
  NP28266 Category 3 | 1
  NP28266 Category 4 | 2

53. Primary Outcome: Number of Participants Who Had Received Mericitabine (MCB)-Based Regimen and Enrolled in NV22688
Description: Population sequencing was used for determination of loss of resistance status. Results are reported as per donor protocol.
Time Frame: Month 18
Population: Resistance monitoring population.
Measure: Number; unit: participants
Groups:
- Resistance Monitoring Arm: Participants enrolled into this arm were those with HCV infection who participated in one of the following donor protocols: NV20536 [NCT00869661], WV21913 [NCT01331850], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], NP28266 [NCT01628094]. None of the enrolled patients had developed MCB-associated resistant mutation(s) in donor protocol. Participants were monitored up to 18 months.
Arm/Group | Resistance Monitoring Arm
Number analyzed (Participants) | 110
participants
  NV20536 | 1
  NV27780 | 2
  NP27946 | 3
  NV27779 | 5
  NP28266 | 6
  WV21913 | 44
  PP25213 | 49

ADVERSE EVENTS:
Time Frame: Up to 36 Months
Description: Only adverse events (AEs) and serious adverse events (SAEs) related to protocol defined blood sampling procedures were collected.
Groups:
- Resistance Monitoring Arm: Participants enrolled into this study were those with Hepatitis C Virus (HCV) infection who participated in one of the following studies (NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094]) and had developed direct acting antiviral (DAA)-associated resistant mutation(s), which persisted through to the last evaluation of drug resistance in the donor protocol(s), or achieved only a partial viral response or experienced a viral breakthrough while on mericitabine treatment not associated with selection of S282T resistance mutations.
- SVR Durability Monitoring Arm: Participants enrolled into this study were those with HCV infection who participated in one of the following studies (NV20536 [NCT00869661], NV21075 [NCT00963885], WV21913 [NCT01331850], NV22621 [NCT01057667], NP22660 [NCT01185860], NV22688 [NCT01168856], NV22776 [NCT01220947], PP25213 [NCT01278134], NV27779 [NCT01482390], NV27780 [NCT01482403], NP27946 [NCT01483742], YV28218 [NCT01749150], NP28266 [NCT01628094]) and had Achieved Sustained Virological Response (SVR-24), defined within the donor protocol as measured by the Roche COBAS TaqMan HCV Test more than or equal to (≥) 20 weeks after the last dose of study medication.
Arm/Group | Resistance Monitoring Arm | SVR Durability Monitoring Arm
Serious Adverse Events (participants affected / at risk) | 0/172 | 0/552
Other Adverse Events (participants affected / at risk) | 1/172 | 0/552
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resistance Monitoring Arm (N=172) | SVR Durability Monitoring Arm (N=552)
VENIPUNCTURE SITE BRUISE (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Investigators were notified of the early termination of study in Jan2015 due to the completion of assessment for resistance monitoring arm and were encouraged to complete scheduled visits until Apr2015 for participants enrolled in SVR durability arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.